CLINICAL TRIAL: NCT05106192
Title: Triamcinolone Acetonide Injections in Primary Cutaneous Lymphoma Plaques With a Novel Needle-free Drug-delivery System.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study closed prior to enrollment of first participant
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE4621
Record Dates: First submitted 2021-10-12; First posted 2021-11-03 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Mycosis Fungoides of Skin (Diagnosis); Cutaneous T-cell Lymphoma; Non Hodgkin Lymphoma; Lymphomatoid Papulosis; Lymphoma, Large-Cell, Anaplastic; Lymphoma, Follicular
MeSH Terms: conditions — Disease; Lymphoma, T-Cell, Cutaneous; Lymphoma, Non-Hodgkin; Lymphomatoid Papulosis; Lymphoma, Large-Cell, Anaplastic; Lymphoma, Follicular | interventions — Triamcinolone Acetonide; Bexarotene; Mechlorethamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Cutaneous T-cell lymphomas (CTCL) Participants (Experimental): The first plaque will be treated using standard of care topical bexarotene or nitrogen mustard for participants with CTCL (cutaneous T-cell lymphomas)
  The second plaque will be treated using a needle-free injector system.
  After the treatment, the participants will be followed for another three visits over the course of 4 months to see how the treated areas responded.
  Interventions: Device: Med-Jet Injector; Drug: Triamcinolone Acetonide; Drug: Bexarotene 1% Top Gel; Drug: Nitrogen Mustard
- Cutaneous B-cell lymphomas (CBCL) Participants (Experimental): The first plaque will be treated using standard of care intralesional TAC (triamcinolone acetonide) using a syringe/needle with participants with CBCL (cutaneous B-cell lymphomas).
  The second plaque will be treated using a needle-free injector system.
  After the treatment, the participants will be followed for another three visits over the course of 4 months to see how the treated areas responded.
  Interventions: Device: Med-Jet Injector; Drug: Triamcinolone Acetonide; Device: Conventional syringe

INTERVENTIONS:
Device: Med-Jet Injector — The Med-Jet injector is a needle-free injection system that consists of a hand-held firing body/trigger, sterilized barrel, disposable luer lock syringe, disposable nozzle cap, and disposable splash guard. The Med-Jet injector is designed to deliver drugs or biologics into the intradermal, subcutaneous, or intramuscular tissues, by means of a narrow, high-velocity jet of fluid, which penetrates the surface of the skin and delivers the fluid to the target tissue
Drug: Triamcinolone Acetonide — The target lesion will be wiped with alcohol and injected with 10mg/ml of TAC directed towards the dermis to create a blanching wheal that is 1 cubic centimeter (total of 0.20 ml of injected fluid).
Drug: Bexarotene 1% Top Gel — Bexarotene can be applied up to four times daily according to patient tolerance directly to lesions. The gel is 1% bexarotene concentration.
  Arms: Cutaneous T-cell lymphomas (CTCL) Participants
Drug: Nitrogen Mustard — Nitrogen mustard is applied once daily as patient tolerates. It is sold in a concentration of 0.016% gel.
  Arms: Cutaneous T-cell lymphomas (CTCL) Participants
Device: Conventional syringe — A standard sterile disposable 1 ml syringe and 30-gauge needle will be used to inject TAC.
  Arms: Cutaneous B-cell lymphomas (CBCL) Participants

SUMMARY:
A study to compare pain differences between using MedJet needle-free drug-delivery system with standard of care treatment for cutaneous T-cell lymphomas and cutaneous B-cell lymphomas in participants.

DETAILED DESCRIPTION:
Participants will undergo treatments on two morphologically and anatomically matched target lesions, preferably on opposing sides of the body.

The first plaque will be treated using standard of care topical bexarotene or nitrogen mustard for participants with CTCL (cutaneous T-cell lymphomas) or intralesional TAC (triamcinolone acetonide) using a syringe/needle with participants with CBCL (cutaneous B-cell lymphomas).

The second plaque will be treated using a needle-free injector system. After the treatment, the participants will be followed for another three visits over the course of 4 months to see how the treated areas responded.

In order to account for 20% dropout, 11 patients per group (a needle free and a traditional treatment group in CBCL patients and the same two groups in CTCL patients) will be recruited.

ELIGIBILITY:
Inclusion Criteria:

1. > 18 years of age
2. Diagnosed with primary cutaneous lymphoma defined by either:

   * A board-certified dermatologist, OR
   * Dermatology Nurse Practitioner, OR
   * Skin punch biopsy
3. The presence of plaque-type primary cutaneous lymphoma lesions with at least two plaques that are at least two cm² in areas of the trunk, buttocks, or extremities that are either:

   * Symmetrically located on contralateral body site OR
   * Within the same body site but separated by ≥ 1 cm
   * Both plaques must be similar in size as much as possible
4. Able to give informed consent under IRB approval procedures

Exclusion Criteria:

1. Known allergy or hypersensitivity to triamcinolone acetonide
2. Known allergy to topical bexarotene or topical nitrogen mustard
3. Pregnant, breastfeeding, or planning to get pregnant 4 weeks before, during, and 4 weeks after the study.
4. Inability to provide informed consent
5. Diagnosis of erythrodermic mycosis fungoides or Sezary syndrome
6. Use of topical corticosteroids to target lesions within 1 week prior to baseline visit
7. Use of radiation therapy to target lesions within 1 week prior to baseline visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Pain measurement between the Med-Jet and standard of care treatment. | 1.5 Hour after the treatment
  The pain of injections with Medjet vs conventional topical therapies of bexarotene or nitrogen mustard will be measured using a visual standard analog pain scale 0 (no distress) to 10 (unbearable distress) immediately after each injection.

SECONDARY OUTCOMES:
Participants Preference | 3 Months
  Number of participants that prefer traditional treatment versus MedJet.
Tolerability of Pruritus | At Baseline, 1 month, 2 months, and 3 months
  Tolerability will be measured using Pruritus score assessment in the Medjet and topical therapy cohorts using a visual standard analog itching scale 0 (no itch) to 10 (worst itch imaginable) with the affected plaques at each indicated visit.
Quality of life due to skin conditions | 3 Months
  The quality of life assessment will be done using the Dermatology Life Quality Index survey (DLQI) which will include a series of topics related to the skin condition including symptoms, feelings, effects on daily life, employment or schooling, personal relationships, and treatment.
  Each of the ten (10) questions are scored from 0 to 3, giving a score range from 0 (meaning no impact of skin disease on quality of life) to 30 (meaning maximum impact on quality of life). Resulting scores are as follows: 0-1 = No effect on patient's life, 2-5 = Small effect, 6-10 = Moderate effect, 11-20 = Very large effect, 21-30 = Extremely large effect.
CAILS assessment of clinical efficacy | At Baseline, 1 month, 2 months, and 3 months
  Composite Assessment of Index Lesion Severity (CAILS) is an assessment of individual lesions by the investigator of disease severity at the time of evaluation which can be used to monitor and compare lesions over time. CAILS is a 5-criterion scale ranging from 0 (no evidence) to 8 (severe), incorporating an assessment of the size of the lesion and severity of erythema, scaling, plaque elevation, and hypo- or hyperpigmentation. When making the assessment of severity, the Investigator will score the area with most clearance (ie, have scores of 0) within the treated plaque.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Cooper, MD, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: It will be immediately available upon request at completion of study.